CLINICAL TRIAL: NCT05426902
Title: Utilizing Qualitative and Quantitative Methods to Understand a New Model of Type 1 and 2 Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00102300; KL2TR002554 (NIH)
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLE@Duke (Experimental): Clinic providers in Duke Rheumatology outside of the Duke Lupus Clinic are eligible to participate in the SLE@Duke intervention. Participants complete a baseline survey and training in the Type 1 & 2 SLE Model. They are asked to perform the intervention for all eligible patients over 4 weeks. Patients complete a survey at the end of their clinic visit, and providers complete a survey at the end of the 4 week intervention period. All participating providers were invited to an in-depth interview at the end of the intervention period.
  Interventions: Behavioral: SLE@Duke

INTERVENTIONS:
Behavioral: SLE@Duke — SLE@Duke is a set of tools to implement the Type 1 & 2 SLE Model in a clinical setting. The model includes an Electronic Medical Record (EMR) note template, patient-reported outcome measure, and training on how to discuss Type 1 & 2 SLE.

SUMMARY:
The purpose of this study is to pilot test SLE@Duke, a set of tools to implement the Type 1 & 2 SLE Model in a clinical setting, as well as to gain an in-depth understanding of providers experiences using the intervention during clinic visits with patients with systemic lupus erythematosus.

This record represents Aim 3 of this study.

ELIGIBILITY:
Inclusion Criteria:

* All providers in Duke Rheumatology who practice outside of the Duke Lupus Clinic are eligible.
* Patients are eligible to participate if they have an established diagnosis of SLE and are followed in Duke Rheumatology.
* All patients with a SLE diagnosis will be included in the analysis. SLE diagnosis will be based on an ICD-10 code for SLE (M32.1*, M32.8, M32.9) in the EMR.

Exclusion Criteria:

* New patients will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Eudy, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients provided data for this study via survey and EMR (electronic medical record), but were not considered enrolled.
Groups:
- Providers: Clinic providers in Duke Rheumatology outside of the Duke Lupus Clinic were eligible to participate in the SLE@Duke intervention. Participants completed a baseline survey and training on the Type 1 & 2 SLE Model. They were asked to perform the intervention for all eligible patients over 4 weeks. Patients completed a survey at the end of their clinic visit, and providers completed a survey at the end of the 4-week intervention period. All participating providers were invited to participate in an in-depth interview at the end of the intervention period.
  SLE@Duke: SLE@Duke is a set of tools to implement the Type 1 & 2 SLE Model in a clinical setting. The model includes an Electronic Medical Record (EMR) note template, patient-reported outcome measure, and training on how to discuss Type 1 & 2 SLE.
- Patients (Survey): Patients who completed an anonymous survey at the end of their clinic visit during the 4-week baseline period and 4-week intervention period.
- Patients (EMR): Electronic medical records (EMRs) of patients with a return visit and diagnosis of SLE who were seen by a participating rheumatology provider were reviewed for outcomes during the 4-week baseline period, 4-week intervention period, and a 4-week follow-up period starting at 3 months after the intervention period.
Period: Overall Study
Arm/Group | Providers | Patients (Survey) | Patients (EMR)
Started | 16 | 49 | 115
Completed | 16 | 49 | 115
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was not collected on the Patients (Survey) group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Providers | Patients (Survey) | Patients (EMR) | Total
Number analyzed (Participants) | 16 | 0 | 115 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data was not collected on Providers or the Patients (Survey) group.
  years
    number analyzed (Participants) | 0 | 0 | 115 | 115
    (all) |  |  | 48.0 (16.2) | 48 (16.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 8 |  | 95 | 103
  Sex/Gender: Male | 5 |  | 20 | 25
  Sex/Gender: Unknown or Not Reported | 3 |  | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 6 | 6
  Not Hispanic or Latino | 13 |  | 106 | 119
  Unknown or Not Reported | 3 |  | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 4 |  | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 1 |  | 67 | 68
  White | 8 |  | 40 | 48
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 3 |  | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 |  | 115 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients' Rheumatologists Using SLE@Duke
Description: Collected from EMR (electronic medical record). This is a composite measure that includes documentation in the clinic note of any component of SLE@Duke: (1) Type 1 & 2 SLE Model mentioned, (2) dotphrase used, (3) Type 1 & Type 2 PGAs (Physician Global Assessments) scored in note, (4) handout mentioned, (5) Type 2 symptoms discussed, or (6) purple sheet documented.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Patients (EMR) group. 36 patient medical records were reviewed during the 4-week baseline period. 31 patient medical records were reviewed during the 4-week intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients (EMR)
Number analyzed (Participants) | 67
Participants
  Baseline: number analyzed (Participants) | 36
  Baseline | 16
  Intervention period: number analyzed (Participants) | 31
  Intervention period | 30
Statistical Analysis 1: Comparison: Patients (EMR); Baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p < 0.0001, Fisher Exact

2. Primary Outcome: Length of Clinic Visits
Description: Collected from EMR (electronic medical record).
Time Frame: Baseline (month 1), intervention period (month 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients (EMR)
Number analyzed (Participants) | 67
minutes
  Baseline (month 1): number analyzed (Participants) | 36
  Baseline (month 1) | 67.8 (22.4)
  Intervention period (month 2): number analyzed (Participants) | 31
  Intervention period (month 2) | 70.9 (28.8)
Statistical Analysis 1: Comparison: Patients (EMR); Baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.6, t-test, 2 sided

3. Primary Outcome: Change in Physician Satisfaction With Visits With Lupus Patients, as Measured by Provider Survey
Description: Satisfaction was measured on a scale of 1-5, where 1 = never and 5 = always in response to the statement: "After seeing a patient with lupus, I leave the exam room feeling satisfied with the encounter."
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Participants who completed the baseline and follow-up surveys. Only applies to the Providers group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 12
score on a scale | 0.44 (0.73)
Statistical Analysis 1: Comparison: Providers; Baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.2, t-test, 2 sided

4. Primary Outcome: Number of Lupus Patients With Assessment of Type 1 and 2 SLE in Note
Description: Collected from EMR (electronic medical record).
Time Frame: Baseline (month 1), intervention period (month 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients (EMR)
Number analyzed (Participants) | 67
Participants
  Baseline (month 1): number analyzed (Participants) | 36
  Baseline (month 1) | 0
  Intervention period (month 2): number analyzed (Participants) | 31
  Intervention period (month 2) | 27
Statistical Analysis 1: Comparison: Patients (EMR); Baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p < 0.0001, Fisher Exact

5. Primary Outcome: Number of Lupus Patients With Type 2 SLE Treatment in Note
Description: Collected from EMR (electronic medical record).
Time Frame: Baseline (month 1), intervention period (month 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients (EMR)
Number analyzed (Participants) | 67
Participants
  Baseline (month 1): number analyzed (Participants) | 36
  Baseline (month 1) | 5
  Intervention period (month 2): number analyzed (Participants) | 31
  Intervention period (month 2) | 8
Statistical Analysis 1: Comparison: Patients (EMR); Baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.4, Fisher Exact

6. Primary Outcome: Perceived Benefits of SLE@Duke, as Measured by Provider Interviews
Description: In-depth interviews with participating rheumatologists related to the intervention, including acceptability, utility, implementation, integration and practicality of SLE@Duke.
Time Frame: 4 weeks
Population: Only applies to the Providers group. Participants who completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 13
Participants
  Improved conversations with patients | 9
  Improved patient understanding | 8
  Improved quality of care | 7
  Validation of patient experiences | 5

7. Primary Outcome: Perceived Barriers of SLE@Duke, as Measured by Provider Interviews
Description: as for outcome 6
Time Frame: 4 weeks
Population: Only applies to the Providers group. Participants who completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 13
Participants
  Need for more training | 4
  Slows down the clinic visit | 4
  Not seeing a lot of lupus patients | 4
  Need for more information on treating Type 2 SLE | 3
  Staff buy-in | 3

8. Primary Outcome: How SLE@Duke Fit Into Work Flow, as Measured by Provider Interviews
Description: as for outcome 6
Time Frame: 4 weeks
Population: Only applies to the Providers group. Participants who completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 13
Participants
  Staff needed more training | 5
  Providers needed more clinic support staff | 4
  Providers had difficulty getting into a routine because of small lupus population in their clinic | 4
  Providers needed a more systematic way of collecting patient surveys | 3
  No impact on work flow | 4

9. Primary Outcome: Number of Lupus Patients With PRO (Patient-reported Outcomes) in Note
Description: Collected from EMR (electronic medical record).
Time Frame: Intervention period (month 2), month 5
Population: Only applies to the Patients (EMR) group. 31 patient medical records were reviewed during the 4-week intervention period. 48 patient medical records were reviewed during the 4-week 3-month follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients (EMR)
Number analyzed (Participants) | 79
Participants
  Intervention period (month 2): number analyzed (Participants) | 31
  Intervention period (month 2) | 0
  Follow-up (month 5): number analyzed (Participants) | 48
  Follow-up (month 5) | 0

10. Primary Outcome: Difference in Perceived Quality of Visit, as Measured by Patient Survey
Description: Each question pertaining to quality of visit was measured on a scale of 1-5, where 1 = strongly disagree and 5 = strongly agree. Different patients completed the survey at month 1 and month 2. The scores at month 1 were averaged, then subtracted from the average score at month 2.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Patients (Survey) group. 19 patients completed surveys during the 4-week baseline period. 30 different patients completed surveys during the 4-week intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients (Survey)
Number analyzed (Participants) | 49
score on a scale
  I feel good about my medical visit. | 0.1 (0.8)
  My rheumatologist gave me his/her full attention. | 0.06 (0.8)
  I was able to say everything I wanted to say to my rheumatologist. | 0.01 (0.7)
Statistical Analysis 1: Comparison: Patients (Survey); "I feel good about my medical visit" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: Patients (Survey); "My rheumatologist gave me his/her full attention" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.8, t-test, 2 sided
Statistical Analysis 3: Comparison: Patients (Survey); "I was able to say everything I wanted to say to my rheumatologist" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 1.0, t-test, 2 sided

11. Primary Outcome: Discussion of the Type 1 and 2 Model, as Measured by Patient Survey
Description: The patient survey asked patients to respond "Yes" or "No" in response to the statement: "My rheumatologist discussed Type 1 & Type 2 lupus with me today."
Time Frame: Intervention period (month 2)
Population: Only applies to the Patients (Survey) group. Patients who responded to the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients (Survey)
Number analyzed (Participants) | 25
Participants
  Yes | 17
  No | 8

12. Primary Outcome: Difference in Understanding of Lupus Activity & Treatment Plan, as Measured by Patient Survey
Description: Questions pertaining to understanding were measured on a scale of 1-5, where 1 = strongly disagree and 5 = strongly agree. Different patients completed the survey at month 1 and month 2. The scores at month 1 were averaged, then subtracted from the average score at month 2.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to Patients (Survey) group. 19 patients completed surveys during the 4-week baseline period. 30 different patients completed surveys during the 4-week intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients (Survey)
Number analyzed (Participants) | 49
score on a scale
  My rheumatologist and I agreed on how active my lupus was today. | 0.1 (0.8)
  I understand the care recommendations that my doctor or provider gave me today. | 0.1 (0.8)
Statistical Analysis 1: Comparison: Patients (Survey); "My rheumatologist and I agreed on how active my lupus was today" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: Patients (Survey); "I understand the care recommendations that my doctor or provider gave me today" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.8, t-test, 2 sided

13. Primary Outcome: Change in Discussion of the Type 1 and 2 Model, as Measured by Provider Survey
Description: Discussion of the Type 1 & 2 SLE Model was measured on a scale of 1-5, where 1 = "never" and 5 = "always" in response to the statement: "I discuss the Type 1 & 2 SLE Model with the patient."
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Providers group. Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 14
score on a scale | 1.0 (0.8)
Statistical Analysis 1: Comparison: Providers; Baseline vs. Follow-Up; Test type: Superiority; p = 0.02, t-test, 2 sided

14. Primary Outcome: Change in Acceptability of SLE@Duke, as Measured by Provider Survey
Description: Questions pertaining to acceptability of SLE@Duke were measured on a scale of 1-5, where 1 = completely disagree and 5 = completely agree.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Providers group. Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 14
score on a scale
  SLE@Duke meets my approval. | -0.1 (0.6)
  SLE@Duke is appealing to me. | 0.0 (0.6)
  I like SLE@Duke. | -0.2 (0.7)
  I welcome SLE@Duke. | -0.2 (0.7)
Statistical Analysis 1: Comparison: Providers; "SLE@Duke meets my approval" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: Providers; "SLE@Duke is appealing to me" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 1.0, t-test, 2 sided
Statistical Analysis 3: Comparison: Providers; "I like SLE@Duke" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.5, t-test, 2 sided
Statistical Analysis 4: Comparison: Providers; "I welcome SLE@Duke" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.6, t-test, 2 sided

15. Primary Outcome: Change in Appropriateness of SLE@Duke, as Measured by Provider Survey
Description: Questions pertaining to the appropriateness of SLE@Duke were measured on a scale of 1-5, where 1 = completely disagree and 5 = completely agree.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Providers group. Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 14
score on a scale
  SLE@Duke seems fitting. | -0.1 (0.6)
  SLE@Duke seems suitable. | -0.1 (0.6)
  SLE@Duke seems applicable. | 0.0 (0.6)
  SLE@Duke seems like a good match. | 0.0 (0.6)
Statistical Analysis 1: Comparison: Providers; "SLE@Duke seems fitting" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: Providers; "SLE@Duke seems suitable" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 3: Comparison: Providers; "SLE@Duke seems applicable" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 1.0, t-test, 2 sided
Statistical Analysis 4: Comparison: Providers; "SLE@Duke seems like a good match" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 1.0, t-test, 2 sided

16. Primary Outcome: Change in Feasibility of SLE@Duke, as Measured by Provider Survey
Description: Questions concerning feasibility of SLE@Duke were measured on a scale of 1-5, where 1 = completely disagree and 5 = completely agree.
Time Frame: Baseline (month 1), intervention period (month 2)
Population: Only applies to the Providers group. Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers
Number analyzed (Participants) | 14
score on a scale
  SLE@Duke seems implementable. | 0.3 (0.6)
  SLE@Duke seems possible. | 0.3 (0.5)
  SLE@Duke seems doable. | 0.2 (0.5)
  SLE@Duke seems easy to use. | 0.4 (0.9)
Statistical Analysis 1: Comparison: Providers; "SLE@Duke seems implementable" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.3, t-test, 2 sided
Statistical Analysis 2: Comparison: Providers; "SLE@Duke seems possible" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.3, t-test, 2 sided
Statistical Analysis 3: Comparison: Providers; "SLE@Duke seems doable" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.4, t-test, 2 sided
Statistical Analysis 4: Comparison: Providers; "SLE@Duke seems easy to use" at baseline (month 1) vs. intervention period (month 2); Test type: Superiority; p = 0.3, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Providers: Clinic providers in Duke Rheumatology outside of the Duke Lupus Clinic are eligible to participate in the SLE@Duke intervention. Participants complete a baseline survey and training in the Type 1 & 2 SLE Model. They are asked to perform the intervention for all eligible patients over 4 weeks. Patients complete a survey at the end of their clinic visit, and providers complete a survey at the end of the 4 week intervention period. All participating providers were invited to an in-depth interview at the end of the intervention period.
  SLE@Duke: SLE@Duke is a set of tools to implement the Type 1 & 2 SLE Model in a clinical setting. The model includes an Electronic Medical Record (EMR) note template, patient-reported outcome measure, and training on how to discuss Type 1 & 2 SLE.
- Patients (EMR): Electronic medical records (EMRs) of patients with a return visit and diagnosis of SLE who were seen by a participating rheumatology provider were reviewed for outcomes during the 4-week baseline period, 4-week intervention period, and 3-month follow-up.
Arm/Group | Providers | Patients (Survey) | Patients (EMR)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/49 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/49 | 0/115
Other Adverse Events (participants affected / at risk) | 0/16 | 0/49 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT05426902/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05426902/ICF_000.pdf